CLINICAL TRIAL: NCT00003125
Title: A Pilot Study of Sequential Vaccinations With ALVAC-CEA and Vaccinia-CEA With the Addition of IL-2 and GM-CSF in Patients With CEA Expressing Tumors
Brief Title: Vaccine Therapy, Interleukin-2, and Sargramostim in Treating Patients With Advanced Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Marshall, MD, Georgetown University
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065885; U01CA062500 (NIH); P30CA051008 (NIH); GUMC-97118; NCI-T97-0033
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer; Esophageal Cancer; Gastric Cancer; Lung Cancer; Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage III gastric cancer; stage IV gastric cancer; stage IIIB breast cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage II esophageal cancer; stage III esophageal cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; unspecified adult solid tumor, protocol specific; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — ALVAC-CEA vaccine; aldesleukin; sargramostim; vaccinia-CEA vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: ALVAC-CEA vaccine
Biological: aldesleukin
Biological: sargramostim
Biological: vaccinia-CEA vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining vaccine therapy, sargramostim, and interleukin-2 may kill more cancer cells.

PURPOSE: Randomized phase II trial to study the effectiveness of vaccine therapy, sargramostim, and interleukin-2 in treating patients who have advanced tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety of sequentially administered vaccinia-carcinoembryonic antigen (CEA) vaccine and ALVAC-CEA vaccine (CEA-Avipox vaccine) in two schedules and with the addition of sargramostim (GM-CSF) plus or minus interleukin-2 (IL-2) in patients with CEA expressing tumors. II. Compare the CEA-specific cellular immune response in cancer patients randomized to receive a single vaccination with vaccinia-CEA vaccine followed by three boosts with ALVAC-CEA vaccine (V-A-A-A) or the reverse vaccination sequence (A-A-A-V). III. Determine whether the addition of GM-CSF alone or with IL-2 enhances the immune response to sequentially administered vaccinia-CEA vaccine and ALVAC-CEA vaccine. IV. Compare the enzyme linked immunosorbent assay ELISPOT with lymphoproliferative and cytotoxicity assays for measuring CEA-specific T lymphocyte immune response.

OUTLINE: This is two-stage, partially randomized study. In stage one, patients are randomized to arm I or II. Arm I: Patients receive vaccinia-carcinoembryonic antigen (CEA) vaccine intradermally on day 1 of course 1 and ALVAC-CEA vaccine (CEA-Avipox vaccine) intramuscularly (IM) on day 1 of courses 2-4. Each course lasts 28 days. Arm II: Patients receive ALVAC-CEA vaccine (CEA-Avipox vaccine) IM on day 1 of courses 1-3 and vaccinia-CEA vaccine intradermally on day 1 of course 4. Each course lasts 28 days. Patients in arms I and II continue 28-day courses through month 6 and then receive 3-month courses for 2 years in the absence of disease progression or unacceptable toxicity. In stage two, patients are enrolled successively into arms III and IV. Arm III: Patients receive vaccines according to whichever schedule (arm I or II) was found to be superior plus sargramostim (GM-CSF) subcutaneously (SC) on days 1-4 of each course. Each course lasts 28 days. Arm IV: Patients receive vaccines plus GM-CSF as in arm III and interleukin-2 SC once daily on days 7-11 of each course. Each course lasts 28 days. Patients on arms III and IV continue 28-day courses through month 6 and then receive 3-month courses for 2 years in the absence of disease progression or unacceptable toxicity. If 2 or more patients in either arm III or IV experience dose limiting toxicity, accrual into study stops. Otherwise, the best response among the 4 arms is determined and further HLA-A2 positive patients are enrolled into that arm so that a total of 6 HLA-A2 positive patients with advanced disease and 6 HLA-A2 positive patients with NED (without radiographic or clinical evidence of tumor) are treated. If more than one regimen is equally superior, the least toxic regimen is chosen for further accrual. Patients are followed at 28 days following the last vaccination.

PROJECTED ACCRUAL: A minimum of 24 patients (6 HLA-A2 positive and up to 3 HLA-A2 negative patients per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignancy that is stage IV and/or at high risk of recurrence despite standard treatment Stage IV malignancy that is surgically rendered free of macroscopic tumor allowed if current available treatment is not likely to offer a survival advantage or result in significant palliation If at high risk for recurrence, must have an estimated recurrence rate of at least 75% following definitive therapy, such as: Postresection of pancreatic cancer Gastric cancer with regional lymph node involvement Node positive stage II or stage III esophageal cancer Stage IIIA or IIIB non-small cell lung cancer Breast cancer with at least 10 positive axillary nodes Must have low tumor burden or no evidence of disease Must have evidence of prior vaccinia (for smallpox immunization) Must have CEA expressing type tumor or a serum CEA elevation of 10 or greater during course of disease No CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: At least 6 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT and SGPT no greater than 4 times ULN Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 50 mL/min Other: HIV negative No uncontrolled seizure disorders, encephalitis, or multiple sclerosis No history of allergy or untoward reaction to prior vaccination with vaccinia virus No other prior or concurrent diagnosis of altered immune function, including eczema, atopic dermatitis, or any autoimmune disease such as systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, Addison's disease, Hashimoto's thyroiditis, or active Graves' disease Must be maintaining a reasonable state of nutrition, consistent with weight maintenance No frequent vomiting or severe anorexia Must be able to avoid close contact with children 3 years or younger, pregnant women, individuals with eczema or history of eczema or other open skin conditions, or immunosuppressed individuals for at least 2 weeks after each vaccination No serious concurrent medical illnesses including inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 6 months after study

PRIOR CONCURRENT THERAPY: Must have recovered from toxic effects of all prior therapy Biologic therapy: Prior vaccinia immunization required No concurrent biologic therapy No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since prior nitrosoureas or mitomycin) No concurrent chemotherapy Endocrine therapy: Physiologic replacement of steroids allowed No concurrent hormonal therapy Radiotherapy: No prior radiotherapy to more than 50% of all nodal groups Surgery: At least 3 weeks since any prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1998-01; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L. Marshall, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - National Naval Medical Center, Bethesda, Maryland